CLINICAL TRIAL: NCT02556632
Title: Effectiveness of Prophylactic Topical Agents for Radiation Dermatitis
Brief Title: Prophylactic Topical Agents in Reducing Radiation-Induced Dermatitis in Patients With Non-inflammatory Breast Cancer
Acronym: Curcumin-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: URCC14079; NCI-2015-00869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC14079 (Other: University of Rochester NCORP Research Base); URCC-14079 (Other: DCP); R21CA178648 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2015-07-23; First posted 2015-09-22 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Carcinoma; Pain; Radiation-Induced Dermatitis; Stage 0 Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Pain; Radiodermatitis; Breast Carcinoma In Situ | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (curcumin-based gel) (Experimental): Patients apply curcumin-based gel topically TID approximately every 4-6 hours beginning on the first day of radiation therapy and continuing until 1 week after completion of radiation therapy.
  Interventions: Drug: Curcumin-based Gel; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm II (HPR Plus) (Experimental): Patients apply HPR Plus™ topically TID approximately every 4-6 hours beginning on the first day of radiation therapy and continuing until 1 week after completion of radiation therapy.
  Interventions: Procedure: Dermatologic Complications Management; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm III (placebo gel) (Placebo Comparator): Patients apply placebo gel topically TID approximately every 4-6 hours beginning on the first day of radiation therapy and continuing until 1 week after completion of radiation therapy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Curcumin-based Gel — Applied topically
  Other Names: Curcumin Gel; Psoria-Gold; Topical Curcumin
  Arms: Arm I (curcumin-based gel)
Procedure: Dermatologic Complications Management — Apply HPR Plus topically
  Arms: Arm II (HPR Plus)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Apply placebo gel topically
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm III (placebo gel)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot phase II trial studies and compares prophylactic topical agents in reducing radiation-induced dermatitis in patients with non-inflammatory breast cancer or breast cancer in situ. The prophylactic topical agents, such as curcumin-based gel or HPR Plus, may reduce the severity of the radiation-induced dermatitis by minimizing water loss and inflammation during radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the effectiveness of Curcumin gel (curcumin-based gel) or HPR Plus™ in reducing radiation dermatitis in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of non-inflammatory breast cancer or carcinoma in situ
* Subjects must be prescribed and scheduled for "conventional fractionated" RT without concurrent chemotherapy; bolus and intensity modulated radiation therapy (IMRT) are permitted; lymph node irradiation (i.e., internal mammary nodes, supraclavicular nodes, axillary nodes, etc) as part of their prescribed radiation therapy are permitted; conventional fractionated radiation therapy regimens eligible for study are described below:

  * Minimal (min) total dose: whole breast: 44 gray (Gy); breast boost: 10 Gy; tumor bed = whole breast +/- boost: 50.0 Gy; lymph nodes: 45 Gy
  * Maximal (max) total dose: whole breast: 50.4 Gy; breast boost: 20 Gy; tumor bed = whole breast +/- boost: 66.0 Gy; lymph nodes: 50.4 Gy
  * Min dose per fraction: whole breast: 1.8 Gy; breast boost: 2.0 Gy; tumor bed = whole breast +/- boost: 1.8 Gy; lymph nodes: 1.8 Gy
  * Max dose per fraction: whole breast: 2.0 Gy; breast boost: 2.0 Gy; tumor bed = whole breast +/- boost: 2.0 Gy; lymph nodes: 2.0 Gy
  * Min # of fractions: whole breast: 22 Gy; breast boost: 5 Gy; tumor bed = whole breast +/- boost: 25 Gy; lymph nodes: 25 Gy
  * Max # of fractions: whole breast: 28 Gy; breast boost: 10 Gy; tumor bed = whole breast +/- boost: 36 Gy; lymph nodes: 28 Gy
  * Min # of sessions: whole breast: 22 Gy; breast boost: 5 Gy; tumor bed = whole breast +/- boost: 25 Gy; lymph nodes: 25 Gy
  * Max # of sessions: whole breast: 28 Gy; breast boost: 10 Gy; tumor bed = whole breast +/- boost: 36 Gy; lymph nodes: 28 Gy
* Subjects may or may not have had surgery (lumpectomy or mastectomy) prior to RT; (NOTE: surgery is not required for eligibility)
* Subjects may have had chemotherapy prior to radiation; a minimum of two weeks is required between end of chemotherapy and start of RT
* Subjects may be currently prescribed hormone treatment or Herceptin therapy
* Subjects must be able to read, speak, and understand English
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Subjects must agree to not use any other topical agents on skin in the radiation treatment area during the course of this trial; subjects should only use topical agents for the study (i.e., topical intervention or standard care agents) supplied by the study personnel and/or treating physician

Exclusion Criteria:

* Pregnant females are ineligible; all subjects of childbearing potential will be asked if they are pregnant or could be pregnant; the patient must respond "no" to continue with radiation and to participate in this clinical study
* Subjects with bilateral breast cancer are not eligible
* Subjects receiving the short-course fractionation radiation therapy (i.e., 16 sessions or 20 sessions at 2.4 to 2.6 Gy fractions per session, with or without boost)
* Subject is currently on anti-EGFR (human epidermal growth factor receptor) therapy, such as Iressa (gefitinib) or Erbitux (cetuximab, C225)
* Previous radiation to the chest or breast
* Subjects with breast reconstruction prior to RT
* Previous diagnosis of radiosensitivity disorder (i.e., ataxia telangiectasia)
* Previous diagnosis of collagen vascular disorder or vasculitis
* Presence of unhealed surgical wounds in chest or breast region and/or breast infection
* Current daily application of a prescribed topical product to the skin within the RT area for an unrelated skin condition that cannot be discontinued during the participation in this clinical trial
* Presence of any active dermatological issues in radiation treatment area (i.e., fungal skin infection, dermatitis, psoriasis plaques, etc)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Morrow, Principal Investigator — University of Rochester NCORP Research Base
Locations (6):
- United States (6):
  - Delaware/Christiana Care NCORP, Newark, Delaware
  - Heartland NCORP, Decatur, Illinois
  - Metro-Minnesota NCORP, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - Columbus NCORP, Columbus, Ohio
  - Dayton Oncology Research Program, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel)
Started | 64 | 65 | 62
Completed | 59 | 59 | 53
Not Completed | 5 | 6 | 9
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Disliked Intervention | 1 | 1 | 1
Not completed — No Reason | 1 | 0 | 1
Not completed — Personal Issues | 0 | 1 | 1
Not completed — Changed Mind | 0 | 1 | 0
Not completed — Withdrew (Unrelated Medical) | 1 | 0 | 0
Not completed — Unrelated Adverse Event | 1 | 0 | 3
Not completed — Related Adverse Event | 0 | 1 | 0
Not completed — Possibly Related Adverse Event | 0 | 0 | 1
Not completed — Did Not Start RT | 0 | 1 | 0
Not completed — Ineligible | 0 | 1 | 0
Not completed — Disliked Study Procedures | 0 | 0 | 1
Not completed — Treatment or Change Delay | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel) | Total
Number analyzed (Participants) | 64 | 65 | 62 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.2) | 60.7 (10.5) | 59.8 (9.3) | 59.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 62 | 191
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 62 | 63 | 61 | 186
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 4 | 21
  White | 55 | 55 | 57 | 167
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Married | 45 | 37 | 37 | 119
  Domestic Partner | 0 | 0 | 1 | 1
  Divorced | 5 | 9 | 16 | 30
  Separated | 1 | 0 | 1 | 2
  Single | 8 | 8 | 2 | 18
  Widowed | 5 | 10 | 4 | 19
  Unknown or Not Reported | 0 | 1 | 1 | 2
Stage of Disease [Count of Participants; unit: Participants] — Ductal carcinoma in situ (DCIS) is considered the earliest form of cancer and consists of abnormal cells in the milk duct.
  Stage I.This stage is a small cancer that has not grown deeply into nearby tissues and has not spread to lymph nodes.
  Stage II and III.These stages indicate larger cancers that have grown more deeply into nearby tissue and may have also spread to lymph nodes.
  Stage IV.This stage means that the cancer has spread to other organs or parts of the body.
  Unknown or Not Reported Stage. There is not enough information to determine stage.
  Participants
    DCIS | 5 | 12 | 11 | 28
    Stage I | 34 | 29 | 22 | 85
    Stage II | 16 | 18 | 20 | 54
    Stage III | 7 | 5 | 8 | 20
    Stage IV | 2 | 0 | 0 | 2
    Unknown or Not Reported | 0 | 1 | 1 | 2
Location of Breast Cancer [Count of Participants; unit: Participants]
  Left | 29 | 27 | 30 | 86
  Right | 35 | 37 | 31 | 103
  Unknown or Not Reported | 0 | 1 | 1 | 2
Prior Chemotherapy [Count of Participants; unit: Participants]
  No | 30 | 35 | 34 | 99
  Yes | 34 | 29 | 27 | 90
  Unknown or Not Reported | 0 | 1 | 1 | 2
Currently on Hormone Therapy [Count of Participants; unit: Participants]
  No | 52 | 48 | 48 | 148
  Yes | 12 | 16 | 13 | 41
  Unknown or Not Reported | 0 | 1 | 1 | 2
Currently on Herceptin Treatment [Count of Participants; unit: Participants]
  No | 56 | 56 | 58 | 170
  Yes | 8 | 8 | 3 | 19
  Unknown or Not Reported | 0 | 1 | 1 | 2
Type of Radiation [Count of Participants; unit: Participants]
  IMRT | 1 | 2 | 2 | 5
  3D Conformal Whole Breast | 63 | 62 | 59 | 184
  Unknown or Not Reported | 0 | 1 | 1 | 2
Radiation Boost Planned [Count of Participants; unit: Participants]
  No | 4 | 3 | 2 | 9
  Yes | 60 | 61 | 59 | 180
  Unknown or Not Reported | 0 | 1 | 1 | 2
Total Radiation Dose Prescribed [Mean (Standard Deviation); unit: Gray units] — The international system (SI) unit of radiation dose expressed in terms of absorbed energy per unit mass of tissue. The gray is the unit of absorbed dose and has replaced the rad. 1 gray = 1 Joule/kilogram and also equals 100 rad. Population: The demographic data was captured in the Onstudy form but two of the participants did not get to the point to fill that form out.
  Gray units
    number analyzed (Participants) | 64 | 64 | 61 | 189
    (all) | 58.4 (5.6) | 59.5 (4.5) | 59.1 (5.2) | 59.0 (5.1)
Breast Field Separation [Mean (Standard Deviation); unit: centimeters] — Breast field separation (BFS) evaluates the association of breast size with radiation-induced skin toxicity. BFS can be obtained from the radiation treatment plan for both 3D conformal breast radiation and IMRT. BFS is defined as the distance between the medial and lateral tangential fields. The tangential fields are created during simulation to achieve uniform dose distribution to the breast volume. The tangential fields align with the medial and lateral contours of the breast. BFS is similar to the width measurement of the breast and is calculated as part of the radiation treatment plan. Population: The demographic data was captured in the Onstudy form but two of the participants did not get to the point to fill that form out.
  centimeters
    number analyzed (Participants) | 64 | 64 | 61 | 189
    (all) | 22.6 (4.0) | 23.8 (4.2) | 22.8 (5.5) | 23.1 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Radiation Dermatitis Severity (RDS) Score. Range: 0 (no Dermatitis) - 4 (Violaceous Erythema With Diffuse Desquamation Occurring in Sheets; Patchy Crusting; Superficial Ulceration)
Description: The mean 1 week post-RT RDS score for each arm will be compared using ANOVA to determine if the topical interventions reduce the severity of skin reactions at the end of RT.
  The RDS score ranges from 0-4 with higher scores indicating worse outcome.
Time Frame: Baseline up to 1 week post radiation therapy
Population: Note: Of the 64 who were randomized to Arm 1, 59 completed the study; of the 65 who were randomized to Arm II, 59 completed the study; of the 62 who were randomized to Arm III, 53 completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel)
Number analyzed (Participants) | 59 | 59 | 53
units on a scale | 2.68 (0.74) | 2.64 (0.74) | 2.63 (0.69)
Statistical Analysis 1: Comparison: Arm I (Curcumin-based Gel) vs Arm II (HPR Plus) vs Arm III (Placebo Gel); Test type: Other; p = 0.9306, ANOVA

2. Primary Outcome: Incidence of Moist Desquamation (Present vs. Absent)
Description: The degree to which each topical intervention decreases the incidence of moist desquamation will be examined using Fisher's exact test. Each agent's potential as a preventative intervention will be determined through comparison of the proportion of subjects with no to minimal radiation dermatitis within each arm using Fisher's exact test.
Time Frame: Baseline up to completion of radiation therapy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel)
Number analyzed (Participants) | 59 | 59 | 53
Participants
  No Moist Desquamation | 44 | 47 | 41
  Moist Desquamation | 15 | 12 | 12
Statistical Analysis 1: Comparison: Arm I (Curcumin-based Gel) vs Arm II (HPR Plus) vs Arm III (Placebo Gel); Test type: Other; p = 0.8048, Fisher Exact

3. Primary Outcome: Change in the Severity of Skin Reactions Using the Radiation Dermatitis Scale (RDS). Range: 0 (no Dermatitis) - 4 (Violaceous Erythema With Diffuse Desquamation Occurring in Sheets; Patchy Crusting; Superficial Ulceration)
Description: The mean 1 week post-RT RDS score for each arm will be compared using ANOVA to determine if the topical interventions reduce the severity of skin reactions after completion of RT.
  The RDS score ranges from 0-4 with higher scores indicating worse outcome.
Time Frame: Baseline to up to 1 week after completion of radiation therapy
Population: Note: Of the 64 who were randomized to Arm 1, 60 completed 1-week post; of the 65 who were randomized to Arm II, 58 completed 1-week post; of the 62 who were randomized to Arm III, 52 completed 1-week post.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel)
Number analyzed (Participants) | 60 | 58 | 52
units on a scale | 2.25 (0.99) | 2.16 (0.92) | 2.15 (0.96)
Statistical Analysis 1: Comparison: Arm I (Curcumin-based Gel) vs Arm II (HPR Plus) vs Arm III (Placebo Gel); Test type: Other; p = 0.8591, ANOVA

ADVERSE EVENTS:
Arm/Group | Arm I (Curcumin-based Gel) | Arm II (HPR Plus) | Arm III (Placebo Gel)
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 3/64 | 2/65 | 6/62
Other Adverse Events (participants affected / at risk) | 8/64 | 3/65 | 5/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Curcumin-based Gel) (N=64) | Arm II (HPR Plus) (N=65) | Arm III (Placebo Gel) (N=62)
Heart Failure (Cardiac disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Radiation Dermatitis (Injury, poisoning and procedural complications) | 3 | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Curcumin-based Gel) (N=64) | Arm II (HPR Plus) (N=65) | Arm III (Placebo Gel) (N=62)
Erythematous papular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Localized edema - Breast swelling (General disorders) | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 1 | 0
Pain (General disorders) | 1 | 1 | 0
Skin and subcutaneous tissue disorders (Other, Specify) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (General disorders) | 0 | 0 | 1
Papulpustular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other: yellow colored bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Vascular disorders - Other: hellow colored hidrosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes